CLINICAL TRIAL: NCT04061499
Title: A Combination of Ultrasound and CT for Investigation of Muscle and Functional Changes in Hip OA Across the Disease Spectrum
Brief Title: Ultrasound and CT to Measure Muscle in Hip OA
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Christa Nelson, Assistant Professor, University of Maryland, Baltimore
Other Study IDs: HP-00087080
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Hip Osteoarthritis
Keywords: muscle; ultrasound; hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hip OA: Individuals with diagnosed hip osteoarthritis
- Control: Individuals without diagnosed hip osteoarthritis

SUMMARY:
This study will examine alterations in muscle in individuals with hip osteoarthritis compared to individuals without hip arthritis. All individuals will receive imaging of their hip and low back muscles in order to compare differences between groups. The investigators hypothesize that there will be differences between groups and that these differences will be related to strength, functional, and balance impairments which will also be measured in all individuals.

DETAILED DESCRIPTION:
Hip osteoarthritis (OA) is one of the most common causes of disability in older adults, with pain, stiffness, and weakness the most frequently reported symptoms. Weakness is a major concern as decreased lower extremity strength is a contributor to balance and other mobility limitations that increase fall risk in the aging population. Weakness in the primary hip muscles in particular have been shown to contribute to gait variability and altered mechanics of stepping when recovering from a balance perturbation. Contributing factors for these strength deficits are multifactorial and may include decreased muscle mass/size, changes in muscle composition, and/or a decreased ability to activate the muscle. Intramuscular fat infiltration (IMAT), has been reported in several conditions affecting older adults, and has been shown to be more modifiable at lower levels, suggesting that earlier detection and intervention may be important. CT and MRI are both commonly used to measure these relevant muscle properties, but ultrasound imaging may be valid alternative, and has the advantage of being more accessible to clinicians in many settings. The investigators hypothesize that cross-sectional area (CSA) and IMAT of the hip and lumbar musculature will be significantly altered in individuals with hip OA (affected limb) compared to that seen in similar-aged control participants, and that larger differences in CSA and IMAT will be positively correlated with OA severity, increased impairment, pain, and disability.

ELIGIBILITY:
Inclusion Criteria:

* Age >=60 and <= 85
* Hip OA group ONLY: Diagnosed unilateral OA of the hip as determined by Kellgren/Lawrence (K/L) or similar grades of 2, 3, or 4 from standard hip series A-P radiographs.
* CONTROL GROUP ONLY: No significant OA of either hip joint as determined by K/L grades or similar of 0 or 1 from standard hip series A-P radiographs.

Exclusion Criteria:

* BMI>35
* Other significant orthopedic conditions of the hip, pelvis or lumbar spine, including prior trauma or significant surgical procedures (examples: lumbar fusion, fractures with surgical management, hip joint replacement, etc.)
* Diagnosis of any other arthritic conditions other than osteoarthritis (e.g. psoriatic arthritis or rheumatoid arthritis, ankylosing spondylitis/spondylosis).
* Any known neurological disorders, including multiple sclerosis, stroke, spinal cord injury or any serious medical condition that may affect muscle quality.
* Inability to undergo CT testing for any reason
* Significant cardiovascular conditions that would make the participant unsafe for any testing procedures (for example uncontrolled hypertension (BP>160/100 at rest), uncontrolled arrhythmia, uncontrolled diabetes, etc.)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Older adults with and without hip osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Muscle cross-sectional area | Day 1
  Muscle CSA will be assessed from CT images and will be reported in units of area, for example square centimeters.
Muscle thickness | Day 1
  Muscle thickness will be assessed from ultrasound images and will be reported in units of length, for example centimeters.
Intramuscular fat infiltration (IMAT) | Day 1
  Assessed from CT images, and measured in Hounsfield units or HU
Echo intensity (EI) | Day 1
  A measure of muscle quality, assessed as the brightness of the ultrasound image using histogram function for each pixel on scale from 0 to 255.

SECONDARY OUTCOMES:
Balance | Day 1
  Balance assessed with Four-square step test
Strength | Day 1
  Muscle strength assessed with Biodex
Mobility | Day 1
  Mobility assessed with Short Physical Performance Battery (SPPB)
Mobility | Day 1
  Mobility assessed with 30-sec chair stand test
Patient self-reported pain and disability: Hip Disability and Osteoarthritis Outcome Score (HOOS) | Day 1
  Hip Disability and Osteoarthritis Outcome Score (HOOS)
  The HOOS is a 40-question questionnaire with five subsections:
  Pain (10 items) Symptoms (5 items) Activities of Daily Living (ADLs - 17 items) Sports and recreations (4 items) Hip-related quality of life (4 items)
  Scoring: Scoring for each question ranges from 0 (never) to extreme (4). A normalized score is calculated for each subscale with 0 representing extreme symptoms and 100 representing no symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Christa Nelson, DPT, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No